CLINICAL TRIAL: NCT03552601
Title: The Effect of Negatively Fluid Balancing Speed for ICU Patients With Acute Respiratory Distress Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Principal Investigator, Bo Yao,phD, Clinician of intensive care unit, Principal Investigator, Qingdao University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YB201806
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Fluid Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional speed (Other): The target amount of every day's net negative fluid balance for the first three days is 1000mL.
  Interventions: Other: traditional speed
- faster speed (Other): The target amount of every day's net negative fluid balance for the first three days is 1500mL.
  Interventions: Other: faster speed

INTERVENTIONS:
Other: traditional speed — ARDS patients are performed negative fluid balance strategy with intravenous furosemide (4mg/h) or continuous veno-venous hemofiltration. The target amount of every day's net negative fluid balance for the first three days is 1000mL.Termination of the strategy is performed when mean arterial pressure drops below 65mmHg or perfusion index drops below 0.82 or lactate increases above 2mmol/L or acute kidney injury occurs.
  Arms: traditional speed
Other: faster speed — ARDS patients are performed negative fluid balance strategy with intravenous furosemide (4mg/h) or continuous veno-venous hemofiltration. The target amount of every day's net negative fluid balance for the first three days is 1500mL.Termination of the strategy is performed when mean arterial pressure drops below 65mmHg or perfusion index drops below 0.82 or lactate increases above 2mmol/L or acute kidney injury occurs.
  Arms: faster speed

SUMMARY:
Previous studies have shown that a positive fluid balance was an independent factor of worse prognosis in ICU patients with acute respiratory distress syndrome (ARDS), and negative fluid balance has been demonstrated to increase oxygenation index, reduce time under mechanical ventilation and ICU length of stay with no noticeable adverse effects. But there is no evidence that faster speed of negative fluid balance would be more beneficial for ARDS patients. So researchers designed the study to prove the effect of negatively fluid balancing speed for ICU patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:

·Patients with ARDS (Berlin 2012 criterion）

Exclusion Criteria:

* Pregnant women
* Unstable hemodynamics status
* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
increased oxygenation index proportion at 24h | at the time of 24 hours
  Oxygenation index equals arterial oxygen partial pressure/fraction of inspiration O2 (PO2/FIO2). Increased oxygenation index proportion at 24h equals (oxygenation index at 24h - oxygenation index at baseline)/ oxygenation index at baseline.

SECONDARY OUTCOMES:
Oxygenation index every day | up to 7 days
  oxygenation index equals arterial oxygen partial pressure/fraction of inspiration O2 (PO2/FIO2).
Duration of free mechanical ventilation | up to 28 days
  Days when patients are free of mechanical ventilation
mortality | up to 28 days
  a measure for the rate at which deaths occur in a given population

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yao, PHD, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The affiliated hospital of qingdao university, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sweeney RM, McAuley DF. Acute respiratory distress syndrome. Lancet. 2016 Nov 12;388(10058):2416-2430. doi: 10.1016/S0140-6736(16)00578-X. Epub 2016 Apr 28. PMID 27133972
- [Result] Sakr Y, Vincent JL, Reinhart K, Groeneveld J, Michalopoulos A, Sprung CL, Artigas A, Ranieri VM; Sepsis Occurence in Acutely Ill Patients Investigators. High tidal volume and positive fluid balance are associated with worse outcome in acute lung injury. Chest. 2005 Nov;128(5):3098-108. doi: 10.1378/chest.128.5.3098. PMID 16304249
- [Result] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Result] Martin GS, Moss M, Wheeler AP, Mealer M, Morris JA, Bernard GR. A randomized, controlled trial of furosemide with or without albumin in hypoproteinemic patients with acute lung injury. Crit Care Med. 2005 Aug;33(8):1681-7. doi: 10.1097/01.ccm.0000171539.47006.02. PMID 16096441
- [Result] Mezidi M, Ould-Chikh M, Deras P, Maury C, Martinez O, Capdevila X, Charbit J. Influence of late fluid management on the outcomes of severe trauma patients: A retrospective analysis of 294 severely-injured patients. Injury. 2017 Sep;48(9):1964-1971. doi: 10.1016/j.injury.2017.06.005. Epub 2017 Jun 15. PMID 28729005
- [Result] Silversides JA, Major E, Ferguson AJ, Mann EE, McAuley DF, Marshall JC, Blackwood B, Fan E. Conservative fluid management or deresuscitation for patients with sepsis or acute respiratory distress syndrome following the resuscitation phase of critical illness: a systematic review and meta-analysis. Intensive Care Med. 2017 Feb;43(2):155-170. doi: 10.1007/s00134-016-4573-3. Epub 2016 Oct 12. PMID 27734109